CLINICAL TRIAL: NCT05029830
Title: Assessment of Quality of Life and Psychological Problems in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samah Ramadan, resident, Assiut University
Other Study IDs: MS
Record Dates: First submitted 2021-06-16; First posted 2021-09-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis Acute and Progressive
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: investigations like MRI.. — • Multiple Sclerosis Quality of Life-54 (MSQOL-54) Can be considered as the most known disease-specific instrument for the evaluation of quality of life in patients with multiple sclerosis (MS). It was developed to combine generic quality of life aspects of the SF-36 with MS-targeted dimensions and ratings for the overall quality of life. Therefore, 18 disease-specific items were added to the original 36 items of the SF-36. The 54 items are divided into 12 multi-item and 2 single-item scales. The MSQOL-54 items are transformed linearly to 0-100 scores and final scores are obtained by averaging items within the scales
  Other Names: questionnaires

SUMMARY:
1. use QoL assessments to check whether interventions have been as effective from the patient's point of view as from the clinician's, and to determine whether further action is required . Knowledge of which factors are determinants of QoL in patients with MS would assist clinicians in choosing the most appropriate interventions. Several determinants of QoL have been identified with varying strengths of association and include both disease-related variables (disability status ,disease duration ,fatigue ,depression ,cognition , sociodemographic variables (age and sex ,level of education, and marital status . A number of these factors might be amenable to treatment intervention, which might be expected to improve QoL: fatigue , depression , and cognition
2. To study effect of psychiatric comorbidity on the disease activity by using clinical, laboratory and psychiometric tools.

DETAILED DESCRIPTION:
2.1 Background (Research Question, Available Data from the literature, Current strategy for dealing with the problem, Rationale of the research that paves the way to the aim(s) of the work). (200-250 words max.) Multiple sclerosis (MS) refers to a chronic, autoimmune and demyelinating inflammatory pathology that affects the Central Nervous System (CNS) in multiple areas, namely the cerebral peduncle and periventricular areas of the brain, optic nerves, and spinal cord . MS is characterized by a diverse set of symptoms and lesions, which can cause serious physical alterations, compromise cognitive functioning, and even trigger neurological problems .

MS etiology is not yet fully understood. However, it is considered a multifactorial disease with environmental and genetic variables being risk factors with immunological implications that alter myelin (white matter) . Myelin, when degraded due to the inflammatory process inherent to the disease (flare-up), can lead to scarring (plaques/lesions) which, in turn, leads to a CNS impairment in the transmission of impulses, resulting in complications in the functioning of several organs.

The impact of MS on patients' quality of life (QoL) is undeniable. However, there are other variables whose influence are significant, such as duration of diagnosis that is associated with worse physical and mental QoL, the degree of disability, and the evolution of the disease, which also appear to be negatively associated with QoL.

Recent studies have attempted to correlate advancing neurologic disability with impaired QOL in MS patients . However, advancing neurologic disability has been shown to only partly explain impaired QOL . This supports the hypothesis that factors other than neurologic disability play a role in the QOL of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* All participants must fulfill the following inclusion criteria: -

  1. fulfillment of either of these five categories of criteria, depending on how many clinical attacks have occurred
  2. patients aged 18 to 40 years of age.
  3. Males and females are included.
  4. All patients who received diagnosis of multiple sclerosis whether under treatment or not.

Exclusion Criteria:

* 1) Patients age of below 18 years or over 40 years . 2) History suggestive or diagnosed collagen disease such as Bechet disease. 3) History suggestive with other general medical disease

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: 1) fulfillment of either of these five categories of criteria, depending on how many clinical attacks have occurred :
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Measurement affection quality of life in patient's with MS | 16 month

SECONDARY OUTCOMES:
Measure psychiatric comorbidity in patients with MS | 16 month

CONTACTS AND LOCATIONS:
Overall Officials: Shady safwat, lecturer, Study Director — Assiut University; gellan karm, lecturer, Study Director — Assiut University
Locations (1):
- Samah, Asyut, Egypt

REFERENCES:
- [Result] Oh J, Vidal-Jordana A, Montalban X. Multiple sclerosis: clinical aspects. Curr Opin Neurol. 2018 Dec;31(6):752-759. doi: 10.1097/WCO.0000000000000622. PMID 30300239